CLINICAL TRIAL: NCT01884064
Title: Multiple Sessions of Low-frequency Repetitive Transcranial Magnetic Stimulation in Focal Hand Dystonia: Clinical and Physiological Effects
Brief Title: Repetitive Transcranial Magnetic Stimulation for the Treatment of Focal Hand Dystonia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Dystonia Medical Research Foundation (Other); National Institutes of Health (NIH) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0608M91226; M01RR000400 (NIH)
Record Dates: First submitted 2012-06-20; First posted 2013-06-21 (Estimated); Results first posted 2015-11-02 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-05

CONDITIONS: Dystonia, Focal, Task-specific
Keywords: focal hand dystonia; rehabilitation; rTMS; writer's cramp; clinical
MeSH Terms: conditions — Dystonia, Focal, Task-Specific; Dystonic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- inhibitory rTMS (Experimental): Repetitive Transcranial Magnetic stimulation: 1 Hz rTMS, 1800 pulses, delivered to premotor cortex. Patients held a pencil and made movements that did not elicit dystonic symptoms during rTMS. Intervention was delivered every day for 5 days.
  Interventions: Device: rTMS
- Sham rTMS (Placebo Comparator): Sham Repetitive Transcranial Magnetic stimulation: 1 Hz rTMS, 1800 pulses, delivered to premotor cortex. Patients held a pencil and made movements that did not elicit dystonic symptoms during rTMS. Intervention was delivered every day for 5 days.
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: rTMS — rTMS
  Other Names: Magstim Rapid 2, Magstim Co, Whitland Dyfed, UK
  Arms: inhibitory rTMS
Device: Sham rTMS — Sham rTMS
  Other Names: Placebo Magstim Rapid 2, Magstim Co, Whitland Dyfed, UK
  Arms: Sham rTMS

SUMMARY:
This study investigated the short term effects of repeated administrations of repetitive-transcranial magnetic stimulation (rTMS) on clinical changes and investigate neurophysiologic responses to rTMS of the activated motor system in patients with FHD.

DETAILED DESCRIPTION:
Purpose: The ability of low-frequency repetitive transcranial magnetic stimulation (rTMS) to enhance intracortical inhibition has motivated its use as a potential therapeutic intervention in focal hand dystonia (FHD). In this preliminary investigation, we assessed the physiologic and behavioral effects of multiple sessions of rTMS in FHD. Methods: 12 patients with FHD underwent five daily-sessions of 1 Hz rTMS to contralateral dorsal premotor cortex (dPMC). Patients held a pencil and made movements that did not elicit dystonic symptoms during rTMS. We hypothesized that an active but non-dystonic motor state would increase beneficial effects of rTMS. Five additional patients received sham-rTMS protocol. The area under curve (AUC) of the motor evoked potentials and the cortical silent period (CSP) were measured to assess changes in corticospinal excitability and intracortical inhibition, respectively. Behavioral measures included pen force and velocity during handwriting and subjective report.

ELIGIBILITY:
Inclusion Criteria:

* Task specific Focal Hand Dystonia

Exclusion Criteria:

* any neurologic condition other than FHD
* medication for dystonia
* botulinum toxin within the past three months
* seizure history
* pregnancy
* implanted medical devices

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa J Kimberley, PhD, PT, Principal Investigator — University of Minnesota
Locations (1):
- Program in Physical Therapy, University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kimberley TJ, Borich MR, Arora S, Siebner HR. Multiple sessions of low-frequency repetitive transcranial magnetic stimulation in focal hand dystonia: clinical and physiological effects. Restor Neurol Neurosci. 2013;31(5):533-42. doi: 10.3233/RNN-120259. PMID 23340117

RESULTS

PARTICIPANT FLOW:
Groups:
- rTMS: Repetitive Transcranial Magnetic stimulation: 1 Hz rTMS, 1800 pulses, delivered to premotor cortex during active hand movement. Intervention was delivered every day for 5 days.
  rTMS: rTMS
- Sham rTMS: Sham or Placebo Repetitive Transcranial Magnetic stimulation: 1 Hz rTMS, 1800 pulses, delivered to premotor cortex during active hand movement. Intervention was delivered every day for 5 days.
  rTMS: rTMS
Period: Overall Study
Arm/Group | rTMS | Sham rTMS
Started | 12 | 5
Completed | 12 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sham rTMS: Sham Repetitive Transcranial Magnetic stimulation: 1 Hz rTMS, 1800 pulses, delivered to premotor cortex during active hand movement. Intervention was delivered every day for 5 days.
  Sham rTMS: Sham rTMS
- Total: Total of all reporting groups
Arm/Group | rTMS | Sham rTMS | Total
Number analyzed (Participants) | 12 | 5 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (12.4) | 46.6 (14.8) | 46.5 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Cortical Silent Period
Description: Subjects performed an isometric abduction contraction of the index finger against a strain gauge coupled to a load cell. A single TMS pulse was applied 2-3 s after contraction initiation and subjects were instructed to relax 2-3 s after stimulation. The duration of the CSP was measured on a trial-by-trial basis and was delineated by the first superimposed TMS-evoked EMG spike (onset) and the return of activity to 50% of prestimulus EMG signal (offset). The mean CSP duration was calculated for each block of measurements. The duration of CSP is thought to be related to intracortical GABAergic synapse-mediated inhibition in the stimulated cortical region. Measures of CSP have been shown to be reliable in repeated measures studies to determine an effect of intervention within a group of subjects (Orth and Rothwell 2004; Borich et al., 2009). Values are calculated as the value recorded at the latest time minus the earliest time point.
Time Frame: Baseline and Day 5
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | rTMS | Sham rTMS
Number analyzed (Participants) | 12 | 5
milliseconds | 9 (6.9) | 1.61 (15.7)

ADVERSE EVENTS:
Time Frame: Before and after each session of the intervention
Description: Subjects were asked to report any adverse event
Arm/Group | rTMS | Sham rTMS
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/5
Other Adverse Events (participants affected / at risk) | 3/12 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rTMS (N=12) | Sham rTMS (N=5)
Mild Headache (Psychiatric disorders) | 2 (2) | 0 (0)
Fatigue (Psychiatric disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
In this preliminary study, there were subjects with different types of hand dystonia and large range of symptom duration. An ideal study would have sufficient n to be able to stratify subjects within various groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No